CLINICAL TRIAL: NCT06820190
Title: Comparison of Analgesic Efficacy of Multiple Mid-Transverse Process to Pleura (MTP) Block and PCA in Idiopathic Scoliosis Patients Undergoing Posterior Spinal Fusion: A Randomized Clinical Trial
Brief Title: Analgesic Efficacy of Multiple Mid-Transverse Process to Pleura (MTP) Block and PCA in Idiopathic Scoliosis Patients Undergoing Posterior Spinal Fusion
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR1047/1/25
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Multiple Mid-Transverse Process to Pleura; PCA; Idiopathic Scoliosis; Posterior Spinal Fusion
MeSH Terms: interventions — Dental Occlusion; Morphine; Passive Cutaneous Anaphylaxis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MTP group (Experimental): Patients will receive multiple mid-transverse process to pleura (MTP) block after induction of anesthesia.
  Interventions: Other: Multiple Mid-Transverse Process to Pleura (MTP) Block
- PCA group (Experimental): Patients will receive IV-PCA. Morphine is generally administered as an initial loading dose of 0.05-0.1 mg/kg before the end of surgery, with PCA settings of a bolus dose of 0.01-0.03 mg/kg, a lockout interval of 6-10 min, and a background infusion of 0.01-0.02 mg/kg/h.
  Interventions: Drug: Morphine

INTERVENTIONS:
Other: Multiple Mid-Transverse Process to Pleura (MTP) Block — Patients will receive multiple mid-transverse process to pleura (MTP) block after induction of anesthesia.
  Arms: MTP group
Drug: Morphine — Patients will receive IV-PCA. Morphine is generally administered as an initial loading dose of 0.05-0.1 mg/kg before the end of surgery, with PCA settings of a bolus dose of 0.01-0.03 mg/kg, a lockout interval of 6-10 min, and a background infusion of 0.01-0.02 mg/kg/h.
  Other Names: PCA
  Arms: PCA group

SUMMARY:
This study aims to compare the analgesic efficacy of multiple mid-transverse process to pleura (MTP) block and PCA in idiopathic scoliosis patients undergoing posterior spinal fusion surgery.

DETAILED DESCRIPTION:
The postoperative period for idiopathic scoliosis patients undergoing posterior spinal fusion (PSF) is fraught with challenges, including adequate postoperative pain control and prolonged hospitalization.

Regional anesthesia techniques, mainly epidural analgesia and, more recently, paravertebral blocks, became crucial parts of the multimodal analgesia (MMA) regimen after introducing ultrasound (US) in the regional anesthesia practice. Erector spinae plane (ESP) block and mid-transverse to pleura (MTP) block are the latest developments in postoperative pain therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years.
* Both sexes.
* American Society of Anesthesiology (ASA) physical status I-II.
* Idiopathic scoliosis patients undergoing posterior spinal fusion surgery.

Exclusion Criteria:

* Patients with pre-existing infection at block site.
* Known allergy to study drugs.
* Coagulation disorder.
* History of psychiatric illness.
* Pre-existing neurological deficits.
* Patient with morbid obesity (body mass index >40 kg/m2).
* Presence of any pre-operative pain or history of chronic pain.
* History of regular analgesic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-02-12 (Actual); Primary Completion 2026-12-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Degree of pain | 24 hours postoperatively
  The degree of pain will be assessed using the Visual Analogue Scale (VAS). VAS (0 represents "no pain" while 10 represents "the worst pain imaginable"). VAS will be assessed at 0, 4, 8, 12, 18 and 24h postoperatively.

SECONDARY OUTCOMES:
Intraoperative fentanyl consumption | Intraoperatively
  Additional fentanyl bolus dosages of 1 µg/kg IV will be administered if heart rate or mean arterial blood pressure elevated more than 20% of the baseline (after exclusion of other causes than pain).
Time to the first request for the rescue analgesia | 24 hours postoperatively
  Time to the first request for the rescue analgesia (time from end of surgery to first dose of morphine administrated).
Total morphine consumption | 24 hours postoperatively
  Postoperative analgesia was provided by morphine (3 mg IV in Multiple Mid-Transverse Process to Pleura (MTP) Block group or 0.01 mg/kg bolus with a 15-min lockout in PCA group) to keep the Visual Analogue Scale (VAS) at rest less than 4.
Mean arterial pressure | Every 15 minutes until the end of the surgery (Up to 2 hours)
  Mean arterial pressure will be recorded preoperatively, before the block is performed, and every 15 minutes until the end of the surgery.
Heart rate | Every 15 minutes until the end of the surgery (Up to 2 hours)
  Heart rate will be recorded preoperatively, before the block is performed, and every 15 minutes until the end of the surgery.
Degree of patient satisfaction | 24 hours postoperatively
  Degree of patient satisfaction will be assessed on a 5-point Likert scale patient satisfaction (1, extremely dissatisfied; 2, unsatisfied; 3, neutral; 4, satisfied; 5, extremely satisfied). It will be assessed 24 hours after surgery.
Incidence of complications | 24 hours postoperatively
  Incidence of complications such as bradycardia, hypotension, nausea, vomiting, Pruritis, respiratory depression, or any other complication will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.